CLINICAL TRIAL: NCT04084080
Title: Sickle Cell Disease and CardiovAscular Risk - Red Cell Exchange Trial (SCD-CARRE)
Acronym: SCD-CARRE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Gladwin, Vice President for Medical Affairs, University of Maryland and Dean, University of Maryland School of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20110362; UG3HL143192 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2019-09-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Erythrocyte Count; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exchange transfusion plus standard of care (Experimental): Randomized to standard of care and automated exchange blood transfusion every 3-6 weeks for 12 months.
  Interventions: Biological: Red Blood Cell; Other: Standard of care
- Standard of care (Active Comparator): Randomized to standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Biological: Red Blood Cell — Red blood cell exchange transfusions will be performed every 3-6 weeks to maintain a target post-transfusion hemoglobin S level of <20% and a pre-transfusion hemoglobin S of <30%.
  Other Names: Red blood cell (RBC)
  Arms: Exchange transfusion plus standard of care
Other: Standard of care — NHLBI/ASH/ATS Expert Panel recommended guidelines

SUMMARY:
The SCD-CARRE trial is a Phase 3, prospective, randomized, multicenter, controlled, parallel two-arm study aimed to determine if automated exchange blood transfusion and standard of care administered to high mortality risk adult SCD patients reduces the total number of episodes of clinical worsening of SCD requiring acute health care encounters (non-elective infusion center/ER/hospital visits) or resulting in death over 12 months as compared with standard of care.

DETAILED DESCRIPTION:
As patients with sickle cell disease (SCD) live to adulthood, the chronic impact of sustained hemolytic anemia and episodic vaso-occlusive events take their toll, with the progressive development of cardiopulmonary organ dysfunction. This culminates in the development of pulmonary hypertension, left ventricular diastolic heart disease, dysrhythmia, chronic kidney disease and sudden death, all major cardiovascular complications of SCD for which there are no approved or consensus therapies. The risk of having pulmonary hypertension and diastolic heart disease can be non-invasively assessed by laboratory tests (NT-proBNP) and Doppler-echocardiography (estimated pulmonary artery systolic pressure). A recent meta-analysis of approximately 6000 patients with SCD demonstrated that patients with elevated tricuspid regurgitant jet velocity (TRV), which is an Doppler-echocardiographic measurement that estimates the pulmonary artery systolic pressure, walked an estimated 30.4 meters less in a 6 minute walk test than those without elevated TRV, and elevated TRV was associated with high mortality (hazard ratio of 4.9). In two large registry cohorts of adult patients with SCD, the investigators found that approximately 20% of the adult SCD population have high values for both biomarkers, defined as a TRV ≥ 2.5 meters per second AND a NT-proBNP ≥ 160 pg/mL, and that the 12-month mortality rate is 7.9% in this group as compared to 0.5% in patients with normal TRV or NT-proBNP values, with a risk ratio for hospitalization of 1.6. This suggests that a simple screening profile of TRV and NT-proBNP can identify about 20% of patients with SCD at the highest risk of death and hospitalization.

Given the increased mortality and early loss of functional capacity associated with cardiovascular disease in SCD adults, it is important to test effective therapeutic interventions in such patients. Red blood cell transfusions are administered by either simple or exchange transfusion, the latter removes the patients blood and replaces it with transfused red blood cells. Exchange transfusions have proven effective for acute treatment of almost all SCD complications, including severe acute chest syndrome, stroke, splenic or hepatic sequestration, and multi-organ failure, and are also used chronically for stroke prevention and recurrent acute chest syndrome. In this study the investigators hypothesize that monthly exchange transfusion will limit disease progression, improve exercise capacity, and prevent interval episodes of vaso-occlusive painful crisis and the acute chest syndrome that acutely increases pulmonary pressures and cause right heart failure.

The investigators propose to perform a clinical trial to evaluate the effects of automated exchange blood transfusion on patient morbidity and mortality, compared to standard of care among 150 adult high risk SCD patients. The trial will leverage existing coordinating center infrastructure at the University of Pittsburgh and will involve 22 experienced clinical sites. Despite the safety and wide utilization of erythrocytapheresis in adult patients with SCD, there is no consensus or quality efficacy data on its use to improve outcomes in our aging high-risk SCD patients with progressive end-organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of SCD: homozygous sickle cell disease, hemoglobin-SC, Sβ-thalassemia, hemoglobin-SO or hemoglobin-SD.
* Patients not on a chronic exchange transfusion program for at least 60 days.
* If patients are on a SCD drug (e.g. hydroxyurea, glutamine, or P-selectin inhibitors), the doses must be stable for at least 60 days prior to randomization. At the time of randomization, participants must be off Oxbryta for at least 30 days.
* Any one of the following vasculopathy biomarker clinical results (a, b, c, d or e) measured in the last 24 months before randomization that indicates a high-risk patient:

  1. Both a TRV 2.5- <3.0 m/sec and NT-proBNP plasma level ≥ 160 pg/mL,
  2. TRV ≥ 3.0 m/sec,
  3. Both a mean pulmonary artery pressure (PAP) by right heart catheterization 20-24 mmHg and NT-proBNP plasma level ≥ 160 pg/mL,
  4. Mean PAP by right heart catheterization ≥ 25 mmHg,
  5. Chronic kidney disease (CKD) due to SCD with abnormal measures on 2 separate occasions as defined by: macroalbuminuria (albumin to creatinine ratio (ACR) >300 mg/g) or proteinuria (protein to creatinine ratio >30 mg/mmol), or estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2. (It is recommended that local laboratories use Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation without ethnic factors when estimating and reporting GFR).

Clinical results of these biomarkers measured locally at sites within 24 months prior to randomization are acceptable to determine eligibility. TRV, PAP, NT-proBNP, albumin to creatinine ratio, protein to creatinine ratio, or eGFR values must be measured in a steady state (defined as measured ≥ 14 days since an acute care pain event) on different days.

vi. Written informed consent obtained from patient to participate in the trial.

Exclusion Criteria:

* RBC alloimmunization resulting in inability of blood bank to obtain compatible components for chronic exchange transfusions
* Previous history of hyper-hemolysis syndrome
* Previous history of severe transfusion reaction resulting in renal failure or due to serious complications such as hypotension or respiratory distress
* More than 10 vaso-occlusive episodes in the past 12 months requiring admission to a hospital to receive treatment.
* Religious objection to receiving blood transfusion
* Diagnosis of ischemic stroke within the past 6 months
* Clinical evidence of liver failure or advanced cirrhosis or any co-existing medical condition that in the Investigator's judgement will substantially increase the risk associated with the patient's participation in the trial
* Women of childbearing potential who have a positive pregnancy test at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Episodes of clinical worsening | 13 months
  The efficacy of the intervention will be measured by comparing the total number of episodes of clinical worsening of SCD requiring acute health care encounters (non-elective infusion center/ER/Hospital visits) or resulting in death over 13 months between groups.

SECONDARY OUTCOMES:
Acute healthcare event | 13 months
  A 6-level prioritized rank-based outcome: 1.No death or SCD-related acute health care encounters (SCDAcuteE) within (w/in) 13 months (m) of randomization; 2. Had SCDAcuteE but NO major complications (acute kidney injury (AKI), acute chest syndrome (ACS), cor pulmonale, stroke, liver failure) associated with an SCDAcuteE nor death w/in 13 m of randomization; 3. Had 1 major complication (AKI, ACS, cor pulmonale, stroke, or liver failure) associated with an SCDAcuteE but not death w/in 13 m of randomization; 4. Had 2 major complications (AKI, ACS, cor pulmonale, stroke, or liver failure) associated with SCDAcuteE but not death w/in 13 m of randomization; 5. Had ≥ 3 major complications (AKI, ACS, cor pulmonale, stroke, or liver failure) associated with SCDAcuteE but not death w/in 13 m of randomization; 6.Death w/in 13 m of randomization. If the same complication reoccurs, occurrences will be counted as separate complications if the acute health care encounters are separated by ≥7 days.
Twelve-month survival | 13 months
  Survival over thirteen-month period will be analyzed and compared between the group receiving the intervention and the group receiving care routinely provided for sickle cell patients based on the NHLBI guidelines.
Survival free of acute healthcare encounters | 13 months
  Survival free of acute health care encounters over 13 months.
Total number of acute health care encounters | 13 months
  The total number of acute health care encounters (non-elective infusion center/ER/Hospital visits) with evidence of cor pulmonale (physical exam findings, NT-proBNP increase plus echocardiographic evidence of worsening right heart function).
Measures of exercise capacity - 6 minute walk distance | 4, 8, and 12 months
  Measures of exercise capacity assessed at 4, 8 and 12 months by the distance walked in the six minute walk distance assessment
Measures of exercise capacity - outpatient activity | 4, 8, and 12 months
  Measures of exercise capacity assessed at 4, 8 and 12 months by the distance walked in a 7 day in the outpatient setting.
Cardiovascular risk | 12 months
  Established cardiovascular risk biomarkers and indices are combined to help the investigators form an opinion about cardiovascular risks. The following will be measured: NT-proBNP, QT prolongation, systemic pulse pressure, albuminuria, estimated GFR and CKD progression Kidney Disease Improving Global Outcomes (KDIGO) CKD Work Group criteria.
Development of new leg ulcers | 4, 8 and 12 months
  Participants will be assessed for development of new leg ulcers at each physical exam.
Measures of exercise capacity - WHO Classification | 4, 8 and 12 months
  WHO functional status severity will be measured assessing by looking at limitation of usual physical activity from I (no limitation in usual physical activity) to Class IV (inability to perform any physical activity at rest)
Nocturnal desaturation | 4, 8 and 12 months
  Nocturnal desaturation will measured using a wearable device to measure blood oxygen saturation for 7 nights at home.
SCD specific patient reported outcomes - Pain | 4, 8 and 12 months
  SCD specific patient reported outcomes as measured by self-reported pain
SCD specific patient reported outcomes -Quality of Life modified PROMIS scale | 4, 8 and 12 months
  SCD specific patient reported outcomes as measured by a modified version of health related quality of life questionnaire from PROMIS QoL measure
SCD specific patient reported outcomes -Quality of Life modified ASCQ-Me scale | 4, 8 and 12 months
  SCD specific patient reported outcomes as measured by a modified version of health related quality of life questionnaire from ASCQ-Me QoL measure
Cardiovascular function by echocardiography - TRV | 4, 8 and 12 months
  Cardiovascular function measures from echocardiography assessed at 4, 8 and 12 months: echocardiographic measures of tricuspid regurgitant jet velocity in m/s.
Cardiovascular function by echocardiography - diastolic left heart function | 4, 8 and 12 months
  Diastolic left heart function measured by E/A ratio, E/Em ratio, and deceleration times will be assessed by echocardiography.
Cardiovascular function by echocardiography - systolic right heart function | 4, 8 and 12 months
  Systolic right heart health will be measured by assessing tricuspid annular plane systolic excursion (TAPSE), right ventricular size and contractility from echocardiography of the heart.
Total number of acute health care encounters | 13 months
  The number of acute health care encounters (non-elective infusion center/ER/Hospital visits) with at least one major complication.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gladwin, MD, Study Chair — University of Maryland; Darrell Triulzi, MD, Principal Investigator — University of Pittsburgh; Maria Brooks, PhD, Principal Investigator — University of Pittsburgh
Locations (23):
- United States (20):
  - University of Alabama, Tuscaloosa, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Howard University Center for Sickle Cell Disease, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Washington University-St. Louis, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Hemorio, Rio de Janeiro, Brazil
- France (2):
  - Kremlin-Bicêtre, Créteil
  - Henri Mondor Hopital, Paris

IPD SHARING:
Plan to Share IPD: Yes
Results from research conducted under this project will be shared in several ways. Manuscripts will be submitted for publication in high-quality peer-reviewed journals, following the NIH Public Access Policy guidelines. Findings will be presented at relevant national conferences, public lectures, scientific institutions and meetings. The timeline for participant recruitment, data collection and analysis will foster publication, facilitated by the investigators' Publications Committee, of critically important and clinically relevant data throughout the trial. The study datasets will be archived and made available to qualified individuals after a period of exclusive use by the SCD-CARRE trial research team and after publication of the primary manuscripts, following NIH guidelines.
Supporting Information: CSR
Time Frame: At the end of the trial, study de-identified datasets will be submitted for permanent archive in the NHLBI BioLINCC repository. The trial will also produce deliverables that will be freely available to the sickle cell community including a description of the protocol for automated red blood cell exchange transfusion.
Access Criteria: All publications based on the SCD-CARRE trial will adhere to the NIH Public Access Policy (Notice NOT-OD-08-033). All study data will be de-identified. At the end of the trial, study de-identified datasets will be submitted for permanent archive in the NHLBI BioLINCC repository.
  The investigators also will work closely with regional and National SCD Foundations to promote recruitment for this study and communicate our results.

REFERENCES:
- [Derived] Abbasi M, Srivastava A, Saraf SL. Management of Kidney Disease with Sickle Cell Disease. J Am Soc Nephrol. 2025 Oct 1;36(10):2041-2054. doi: 10.1681/ASN.0000000804. Epub 2025 Jun 26. PMID 40569673